CLINICAL TRIAL: NCT07308158
Title: Human Factors and Clinical Validation of the iHealth Labs Inc iHealth Flu A&B/COVID-19/RSV Rapid Test in Anterior Nares Nasal Samples For Over the Counter (OTC) Use
Brief Title: Covid Flu A/B and RSV 4 in 1 Diagnostic Test
Status: Completed | Type: Observational
Sponsor: iHealth Labs inc (Industry)
Responsible Party: Sponsor
Other Study IDs: iH018
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Influenza A; Influenza B; COVID - 19; RSV
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Investigational Flu A/B Covid-19 and RSV Diagnostic Test — A diagnostic test in lateral flow cassette format designed to detect Influenza A, Influenza B, SARS-CoV-2 and respiratory syncytial virus from anterior nasal swab specimens.

SUMMARY:
The goal of this observational study is to evaluate the diagnostic performance of an investigational Flu A/B, COVID-19 and RSV test in patients with signs and symptoms of respiratory infection.

The main questions it aims to answer are:

1. What is the sensitivity and specificity of the investigational test compared with an FDA-cleared reference method for detection of Influenza A, Influenza B, , SARS-CoV-2 and respiratory syncytial virus antigen.
2. What is the overall positive and negative percent agreement between the investigational test and the reference method?

Participants will:

1. Provide a respiratory specimen (e.g., nasal or nasopharyngeal swab) for testing with the investigational device.
2. Provide an additional specimen for testing with the FDA-cleared reference method.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to study enrollment.
* Male or female aged six (6) months or older.
* Subject is currently exhibiting two or more symptoms associated with COVID-19, influenza or RSV (such as, but not limited to, fever, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting or diarrhea and must present within six (6) days of symptom onset). Subject must still be exhibiting symptoms on the day of sample collection.

Exclusion Criteria:

* Subject who is 18 years of age (or the state's legal age of majority) or older and does not understand or is not able and willing to sign the study informed consent.
* Subject has had seasonal influenza and/or the SARS-CoV-2 and/or the RSV vaccine within the past 5 days.
* Subject is not able to tolerate sample collection, or is not willing to contribute the required swab samples for testing or complete the study procedures.
* Subject is currently undergoing antiviral treatment such as baloxavir marboxil (trade name Xofluza®), oseltamivir (Tamiflu®), zanamivir (Relenza®), or peramivir (Rapivab®).
* Subjects currently undergoing treatment and/or within the past thirty (30) days with prescription medication to treat novel Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury), Paxlovid, molnupiravir or receiving convalescent plasma therapy for SARS-CoV-2.
* Subjects who have taken Evusheld (tixagevimab/cilgavimab) within the last 90 days.
* Subjects who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to the study sample collection.
* Subjects who have had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with flu-like symptoms presenting to participating clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 1119 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Investigational Test for Detection of Influenza A, Influenza B, SARS-CoV-2 and Respiratory Syncytial Virus Compared to an FDA-Cleared Reference Method | Within approximately 5 days of specimen collection (time needed for both investigational and comparator test results)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (21):
  - iHealth Site 006, Birmingham, Alabama
  - iHealth Site 021, Trussville, Alabama
  - iHealth Site 017, Dublin, California
  - iHealth Site 007, Huntington Park, California
  - iHealth Site 026, Toluca Lake, California
  - iHealth Site 011, DeLand, Florida
  - iHealth Site 013, Doral, Florida
  - iHealth Site 004, Fort Lauderdale, Florida
  - iHealth Site 005, Fort Lauderdale, Florida
  - iHealth Site 019, Palm Springs, Florida
  - iHealth Site 014, Tamarac, Florida
  - iHealth Site 009, Ammon, Idaho
  - iHealth Site 027, Edison, New Jersey
  - iHealth Site 015, Simpsonville, South Carolina
  - iHealth Site 016, Spartanburg, South Carolina
  - iHealth Site 020, Chattanooga, Tennessee
  - iHealth Site 003, Brownsville, Texas
  - iHealth Site 002, Edinburg, Texas
  - iHealth Site 018, El Paso, Texas
  - iHealth Site 023, Mesquite, Texas
  - iHealth Site 025, Morgantown, West Virginia
- Puerto Rico (2):
  - iHealth Site 001, Quebradillas
  - iHealth Site 022, San Juan

IPD SHARING:
Plan to Share IPD: No